CLINICAL TRIAL: NCT02571114
Title: A Randomized, Controlled Study to Examine the Glycemic and Metabolic Responses of Frozen Yogurt Containing Saskatoon Berry Powder in Healthy Males and Females
Brief Title: Glycemic and Metabolic Responses of Frozen Yogurt Containing Saskatoon Berry Powder in Healthy Males and Females
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: B2014:121
Record Dates: First submitted 2015-10-06; First posted 2015-10-08 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-09

CONDITIONS: Healthy
Keywords: Glycemic Responses; Metabolic Responses; Males; Females

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Control 1 (Active Comparator): white bread - 25 g available carbohydrate
  Interventions: Dietary Supplement: Control 1
- Control 2 (Active Comparator): white bread - 25 g available carbohydrate
  Interventions: Dietary Supplement: Control 2
- Frozen Yogurt (Sham Comparator): unflavoured frozen yogurt - 25 g available carbohydrate
  Interventions: Dietary Supplement: Frozen Yogurt
- Saskatoon Berry Frozen Yogurt (Experimental): frozen yogurt containing powder prepared from Saskatoon berries - 25 g available carbohydrate
  Interventions: Dietary Supplement: Saskatoon Berry Frozen Yogurt

INTERVENTIONS:
Dietary Supplement: Saskatoon Berry Frozen Yogurt — Frozen yogurt containing a defined amount of powder prepared from Saskatoon berries (serving size = 25 g available carbohydrate)
  Arms: Saskatoon Berry Frozen Yogurt
Dietary Supplement: Frozen Yogurt — Unflavoured frozen yogurt (serving size = 25 g available carbohydrate)
  Arms: Frozen Yogurt
Dietary Supplement: Control 1 — White bread (serving size = 25 g available carbohydrate)
  Arms: Control 1
Dietary Supplement: Control 2 — White bread (serving size = 25 g available carbohydrate)
  Arms: Control 2

SUMMARY:
A single site, blinded, randomized, controlled study designed to examine the glycemic and metabolic response of frozen yogurt containing Saskatoon berry powder in healthy males and females.

DETAILED DESCRIPTION:
A single site, blinded, randomized, controlled study designed to examine the glycemic and metabolic response of frozen yogurt containing Saskatoon berry powder in healthy males and females. Eligible participants will be asked to attend 4 in-person clinic visits for comparative testing of the frozen yogurt and frozen yogurt containing Saskatoon berry powder versus white bread. Separate visits for screening and for a fasting blood sample will also be requested (total of 6 visits).

ELIGIBILITY:
Inclusion Criteria:

1. Male, or non-pregnant, non-lactating female, ≥18 and ≤35 years;
2. Normal blood lipid profile, creatinine <1.5× upper limit of normal (ULN) where the normal range is ≥7 units/L and ≤56 units/L, alanine aminotransferase (ALT) <2× ULN where the normal range is ≥0.7 mg/dL and ≤1.3 mg/dL, and glycated hemoglobin <6%;
3. Blood pressure <140/90
4. Body mass index (BMI) ≥20 and <30;
5. Stable regime for the past 3 months if taking vitamin and mineral/dietary/ herbal supplements;
6. Agree not to eat Saskatoon berries or foods containing Saskatoon berries while participating in this study;
7. Willing to comply with the protocol requirements;
8. Willing to provide informed consent.

Exclusion Criteria:

1. Not able to consume yogurt or allergies to Saskatoon berries or ingredients in yogurt or bread;
2. Presence of a clinically diagnosed disease affecting the circulatory, respiratory, immune, skeletal, urinary, muscular, endocrine, digestive, nervous or reproductive system that requires medical treatment;
3. Taking any prescribed medication in the last 3 months or supplements that affect gastrointestinal function in the last 3 months;
4. Weight loss of ≥3 kg of body weight within the 6 months prior to enrolling in the study;
5. Current (within the last month) bacterial, viral or fungal infection, or over-the-counter medication within the past 72 hours;
6. Unable to obtain blood samples at the screening or the first study visit.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2015-10; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Serum glucose | 180 min
  glucometer readings of serum glucose at intervals after consumption of study foods

SECONDARY OUTCOMES:
serum insulin | 180 min
  serum insulin levels in response to consumption of study foods
metabolomics | 180 min
  mass spectrometry analysis of serum and urine before and after consumption of study foods

CONTACTS AND LOCATIONS:
Overall Officials: Carla G Taylor, PhD, Principal Investigator — St. Boniface Hospital Asper Clinical Research Institute
Locations (1):
- St. Boniface Hospital, Asper Clinical Research Institute, Winnipeg, Manitoba, Canada

REFERENCES:
- [Derived] Pauls SD, Du Y, Clair L, Winter T, Aukema HM, Taylor CG, Zahradka P. Impact of Age, Menopause, and Obesity on Oxylipins Linked to Vascular Health. Arterioscler Thromb Vasc Biol. 2021 Feb;41(2):883-897. doi: 10.1161/ATVBAHA.120.315133. Epub 2020 Dec 31. PMID 33380172